CLINICAL TRIAL: NCT02915211
Title: A Feasibility Study to Evaluate the Acceptability of Keyo, a Food for Special Medical Purposes (FSMP) for Use in the Ketogenic Diet (KD) With Regard to Product Tolerance, Compliance and Acceptability
Brief Title: Evaluation of Keyo in Children With Epilepsy
Acronym: Keyo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCT-Keyo-11/12/15-01; 196542 (Other: IRAS)
Record Dates: First submitted 2016-09-19; First posted 2016-09-26 (Estimated); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Intractable Epilepsy; Glucose Transporter Type 1 Deficiency Syndrome; Ketogenic Dieting
Keywords: Epilepsy; Glut; Ketogenic; Glucose
MeSH Terms: conditions — Drug Resistant Epilepsy; Glut1 Deficiency Syndrome; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Consumption of Keyo (Experimental): Participants will consume their normal KD and take Keyo as advised by the lead dietitian.
  Interventions: Dietary Supplement: Keyo

INTERVENTIONS:
Dietary Supplement: Keyo — Keyo is a Food for Special Medical Purposes (FSMP) and is intended for use in the KD. It has a fat to protein and carbohydrate ratio of 3 to 1. This makes it appropriate for inclusion in all versions of the KD - classical, MCT, MAD and LGI. Keyo has been designed as a nutritionally complete, ready to use, pleasant tasting and versatile medical food for use in a KD.

SUMMARY:
To evaluate the tolerance, acceptability and compliance of Keyo in 20 subjects aged 3 years and over, with intractable epilepsy or Glut-1 DS on a KD.

DETAILED DESCRIPTION:
Qualitative assessments from subject questionnaires that allow evaluation of the acceptability and ease of use of the study product.

Collection of daily data about the gastro-intestinal tolerance of the study product.

Collection of daily data about compliance with the study product i.e. actual versus prescribed intake.

Improve quality of life by increasing range of foods available for use in a ketogenic diet.

ELIGIBILITY:
Inclusion Criteria:

* 3 years and over
* Confirmed diagnosis of intractable epilepsy or Glut-1 DS
* Children must be currently established on a KD for at least 3 months, taken orally
* Written, informed consent by participant/carer

Exclusion Criteria:

-

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Palatability questionnaire | Day 8
  Qualitative assessment from subject questionnaire that allows evaluation of the palatability of the study product.
Ease of use daily diary | Days 1-7
  Qualitative assessments from subject questionnaires that allow evaluation of the ease of use of the study product.
GI tolerance daily diary | Days 1-7
  Qualitative assessments from subject questionnaires that allow evaluation of the gastro-intestinal tolerance of the study product.
Product compliance daily diary | Days 1-7
  Qualitative assessments from subject questionnaires that allow evaluation of compliance with the study product, i.e. actual versus prescribed intake.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McCullagh, BSc, MBChB, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (2):
- United Kingdom (2):
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester, Greater Manchester
  - Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: Undecided